CLINICAL TRIAL: NCT04127214
Title: The ITA Model of Integrated Treatment of Eating Disorders
Acronym: ITAMITED
Status: Active, not recruiting | Type: Observational
Sponsor: University of Barcelona (Other)
Collaborators: ITA salud mental (Unknown)
Responsible Party: Principal Investigator, Dr. Guillem Feixas, Professor, University of Barcelona
Other Study IDs: FBG309562
Record Dates: First submitted 2019-10-01; First posted 2019-10-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge Eating; Eating Disorders in Adolescence; Eating and Feeding Disorders
Keywords: eating disorders; anorexia nervosa; bulimia nervosa; binge eating; routine outcome monitoring; psychological interventions; integrated treatment; effectiveness
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Bulimia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ITA Integrated Treatment — The ITA Model combines outpatient intervention (mainly psychotherapy), day hospital care and hospitalization as a function of patients' characteristics. Case conceptualization of the psychological processes of patients is formulated and revised within a team including psychologists, psychotherapists, psychiatrists, nutritionists, physicians, nurses, and social workers. The major emphasis of the ITA model is on psychological interventions which include individual psychotherapy, family therapy and/or guidance, and group therapy of various formats and contents (e.g., drug abuse, mindfulness, emotion work) tailored to the needs of each patient. However, when required, drugs are prescribed adjusting type of medication and dosage to the need of the patient.

SUMMARY:
This is a naturalistic study implementing a routine assessment to monitor the evolution of the patients with eating disorders being treated in various centers of "ITA salud mental" in Spain.

DETAILED DESCRIPTION:
"ITA salud mental" offers integrated treatment for eating disorders including outpatient, inpatient and day hospital care. The routine assessment implemented to this aim includes both general measures to gauge the therapeutic progress (CORE system) and measures specific for eating disorders (EAT, BITE), which are administered from the beginning to the end of treatment in different time points combined with clinical data included in the patients' health record such as diagnosis, body mass index, previous treatments, and chronicity.

According to its naturalistic nature, this study will accept all participants who are admitted into the care system offered by "ITA salud mental" between November 2, 2017 and October, 2nd., 2020, meeting the inclusion/exclusion criteria and signing informed consent (n = 800 is an estimation). These patients will be followed on three-week bases until October, 30th., 2020, and less intensively on three-month bases until October 2025 to monitor symptoms and to record possible adverse effects.

The analysis of these data will permit to evaluate the therapeutic effects of this integrated treatment and the factors which might influence the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an eating disorder: Anorexia Nervosa, Bulimia Nervosa, Binge and other eating disorders Not Otherwise Specified.
* Treated in one of the centers of "ITA salud mental".

Exclusion Criteria:

* Not willing to participate (not signing informed consent).

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with eating disorders undergoing treatment at "ITA salud mental".
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical outcomes in routine evaluation outcome measure (CORE-OM) | CORE-OM is administered at baseline, at one week, and then routinely every three months (using A and B short forms alternatively every three weeks until October 30th, 2020) until study completion.
  CORE-OM is a 34-item self-report questionnaire for the assessment of subjective well-being, symptoms or problems, life functioning, and risk. It has good psychometric properties and it has been validated for the Spanish population. Its transdiagnostic nature makes it suitable for all kinds of eating disorders especially if we take into account the frequent comorbidities with other mental disorders (e.g., depression, anxiety) of these patients. Short forms of this questionnaire (versions A and B) are used to monitor patients' progress.
Change in Eating Attitudes Test (EAT) | EAT is administered at baseline, at one week, and then routinely every three months until study completion.
  The EAT (children and adult versions) is a 26-item standardized self-report questionnaire devised to measure symptoms and concerns characteristic of eating disorders. Although the EAT has been used as a screening tool, here it is used to gauge symptom severity. It has good psychometric properties and it has been validated for the Spanish population.

SECONDARY OUTCOMES:
Change in Bulimic Investigatory Test, Edinburgh (BITE) | BITE is administered at baseline, at one week, and then routinely every three months until 30th. of October, 2020.
  BITE is a 33-item standardized self-report questionnaire measuring eating disorders symptoms and severity. It is especially suited for binge eating disorders and bulimia nervosa. The test is well sensitive to measure the effectiveness of the therapy and the changes of symptoms. It has good psychometric properties and it has been validated for the Spanish population.
Change in Body Mass Index (BMI) | Patients' weight and height is recorded at baseline and then weight every month (every thee-months after October 30th, 2020) up to 5 years. No follow-up data will be collected for this measure.
  The BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in meters. It is widely used for the assessment of therapeutic progress in eating disorders and obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Feixas, PhD, Principal Investigator — Universitat de Barcelona, Spain; Antoni Grau-Touriño, Psychologist, Study Director — ITA salud mental, Spain; Chris Evans, MD, Study Chair — University of Sheffield, UK
Locations (8):
- Spain (8):
  - ITA salud mental-Argentona, Argentona, Catalonia
  - ITA salud mental-Avenir, Barcelona, Catalonia
  - ITA saklud mental-Urgell, Barcelona, Catalonia
  - ITA salud mental-Sabadell, Barcelona, Catalonia
  - ITA saludmental-Tarragona, Tarragona, Catalonia
  - ITA salud mental-Moscatelar, Madrid
  - ITA salud mental-Alcalá, Madrid
  - ITA salud mental-ABB Sevilla Vidrio, Seville

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grau Tourino A, Feixas G, Medina JC, Paz C, Evans C. Effectiveness of integrated treatment for eating disorders in Spain: protocol for a multicentre, naturalistic, observational study. BMJ Open. 2021 Mar 8;11(3):e043152. doi: 10.1136/bmjopen-2020-043152. PMID 34006027
- See also: Research group on Intervention in Clinical and Health Psychology (recognized by the "Generalitat de Catalunya") — http://ub.edu/ipcs
- See also: Web site of "ITA salud mental" the institution in which the study is conducted — http://itasaludmental.com

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT04127214/SAP_000.pdf